CLINICAL TRIAL: NCT07389330
Title: Patients' Perceptions of Postoperative Analgesic Monitoring in Elective General Surgery: A Mixed-Methods Structural Equation Modeling Study
Brief Title: Patients' Perceptions of Postoperative Analgesic Monitoring in Elective General Surgery
Acronym: PSAM-SEM
Status: Not yet recruiting | Type: Observational
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Volkan Gokmen, Assistant Professor, Agri Ibrahim Cecen University
Other Study IDs: PSAM-SEM-2026
Record Dates: First submitted 2026-01-25; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Pain Management
Keywords: postoperative analgesic monitoring; elective general surgery; pain disclosure; trust in nursing care; structural equation modeling
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective General Surgery Patients: Adult patients undergoing elective general surgery who receive routine postoperative analgesic monitoring as part of standard clinical care.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention is applied in this study. Participants receive standard postoperative care, including routine analgesic monitoring, as part of usual clinical practice.

SUMMARY:
This study examines how patients perceive postoperative analgesic monitoring during routine care in elective general surgery. Postoperative pain monitoring is a standard nursing practice, but patients may experience it as either supportive or stressful. These perceptions may influence patients' trust in nursing care, anxiety related to monitoring, and willingness to report pain accurately.

The study uses a mixed-methods observational design. In the quantitative phase, patients complete questionnaires about their experiences with pain monitoring, communication with nurses, trust, anxiety, and pain reporting during the first days after surgery. In the qualitative phase, selected patients participate in interviews to further explain and contextualize the survey findings. No changes are made to standard care, and no experimental treatments are used.

DETAILED DESCRIPTION:
Postoperative analgesic monitoring is a routine component of nursing care in elective general surgery and is essential for patient safety and effective pain management. Although monitoring practices are intended to support patients, they may also be perceived as stressful or controlling, depending on how they are experienced and communicated. These perceptions may influence psychosocial processes such as trust in nursing care, anxiety related to monitoring, and patients' willingness to disclose pain.

This study is designed as a prospective observational mixed-methods study conducted in elective general surgery wards. No intervention is applied, and all participants receive standard postoperative care according to institutional protocols. The quantitative phase involves patient-reported questionnaires administered during the first 72 hours after surgery. These measures assess perceptions of postoperative analgesic monitoring, trust in nursing care, monitoring-related anxiety, pain disclosure behavior, and perceived quality of nursing communication.

Structural equation modeling is used to examine the relationships among these variables and to test hypothesized pathways between monitoring perceptions and pain disclosure behavior. The qualitative phase consists of in-depth interviews with a purposive subsample of participants selected based on contrasting survey responses. These interviews are used to explain and enrich the quantitative findings by exploring patients' experiences and interpretations of analgesic monitoring and communication.

Quantitative and qualitative findings are integrated during interpretation to provide a comprehensive understanding of how postoperative analgesic monitoring is perceived by patients and how these perceptions may influence communication and behavior related to pain management. The study aims to generate evidence that can inform patient-centered approaches to postoperative analgesic monitoring while maintaining routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Undergoing elective general surgery requiring postoperative inpatient care
* Receiving routine postoperative analgesic monitoring as part of standard clinical care
* Clinically stable during the postoperative data collection period
* Able to read and communicate in Turkish
* Able and willing to provide written informed consent

Exclusion Criteria:

* Emergency or urgent surgical procedures
* Postoperative admission to an intensive care unit
* Requirement for mechanical ventilation
* Documented cognitive impairment, acute delirium, or severe psychiatric illness
* Inability or unwillingness to complete study questionnaires or interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing elective general surgery who are hospitalized postoperatively and receive routine analgesic monitoring as part of standard nursing care in a tertiary university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain Disclosure Behavior | Postoperative days 1 to 3
  Pain disclosure behavior is measured using the Pain Disclosure Behavior Scale (PDB), a self-report questionnaire consisting of 3 items. Each item is rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 3 to 15, with higher scores indicating greater willingness to report pain accurately and to request analgesia when needed.

SECONDARY OUTCOMES:
Trust in Nursing Care | Postoperative days 1 to 3
  Trust in nursing care is assessed using the Trust in Nursing Care Scale (TNC), a 3-item self-report instrument. Items are rated on a 5-point Likert scale from 1 (very low trust) to 5 (very high trust). Total scores range from 3 to 15, with higher scores indicating greater trust in nursing competence, intentions, and clinical judgment.
Monitoring-Related Anxiety | Postoperative days 1 to 3
  Monitoring-related anxiety is measured using the Monitoring-Related Anxiety Scale (MRA), a 3-item self-report questionnaire. Each item is scored on a 5-point Likert scale from 1 (not anxious at all) to 5 (extremely anxious). Total scores range from 3 to 15, with higher scores indicating greater anxiety related to postoperative analgesic monitoring.
Perceived Surveillance-Oriented Analgesic Monitoring | Postoperative days 1 to 3
  Perceived surveillance-oriented analgesic monitoring is assessed using the Perceived Surveillance of Analgesic Monitoring Scale (PSAM). The scale consists of 3 items rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 3 to 15, with higher scores reflecting stronger perceptions of monitoring as controlling or surveillance-oriented.
Perceived Supportive Analgesic Monitoring | Postoperative days 1 to 3
  Perceived supportive analgesic monitoring is measured using the Perceived Supportive Monitoring Scale (PSM), a 3-item self-report instrument. Items are scored on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 3 to 15, with higher scores indicating greater perception of analgesic monitoring as supportive and reassuring.
Perceived Nursing Communication Quality | Postoperative days 1 to 3
  Nursing communication quality is assessed using a validated Nursing Communication Quality Scale consisting of 4 items. Each item is rated on a 5-point Likert scale from 1 (very poor communication) to 5 (excellent communication). Total scores range from 4 to 20, with higher scores indicating better perceived communication quality.

OTHER OUTCOMES:
Patient Experiences of Postoperative Analgesic Monitoring | Up to 48 hours following surgery
  Qualitative experiences of postoperative analgesic monitoring are collected through semi-structured interviews. Data are recorded as verbatim textual transcripts and analyzed thematically. No numerical unit of measurement is applied.

CONTACTS AND LOCATIONS:
Locations (1):
- Ağrı Training and Research Hospital, AĞRI, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study involves patient-reported perceptions, psychosocial measures, and qualitative interview data collected in a postoperative clinical setting. Sharing IPD could pose a risk to participant confidentiality and privacy. Only aggregated and anonymized results will be reported in publications.

REFERENCES:
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Salmon P, Manyande A. Good patients cope with their pain: postoperative analgesia and nurses' perceptions of their patients' pain. Pain. 1996 Nov;68(1):63-68. doi: 10.1016/S0304-3959(96)03171-5. PMID 9251999
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Background] Qaddumi J, Arda AM, Alkhawaldeh A, ALBashtawy M, Abdalrahim A, ALBashtawy S, Al Omari O, Bashtawi M, Masa'deh R, ALBashtawy Z, Mohammad KI, ALBashtawy B, Aljezawi M, Khatatbeh H, Ta'an W, Suliman M, Al Dameery K, Bani Hani S. Preoperative anxiety, postoperative pain tolerance and analgesia consumption: A prospective cohort study. J Perioper Pract. 2025 Oct;35(10):426-436. doi: 10.1177/17504589241253489. Epub 2024 Aug 6. PMID 39104294